CLINICAL TRIAL: NCT04264793
Title: Skills for Change: Implementation of a Community-based Diabetes Nutrition Education Program for Emirati Adults With Type 2 Diabetes
Brief Title: Skills for Change: Nutrition Education Program for Emirati Adults With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United Arab Emirates University (Other)
Collaborators: Ambulatory Healthcare Services, Al Ain, UAE (Unknown); Sheikh Hamdan bin Rashid Al Maktoum Award for Medical Sciences (Unknown)
Responsible Party: Principal Investigator, Habiba I. Ali, Associate Professor, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/48
Record Dates: First submitted 2020-02-08; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes
Keywords: Emirati Adults; United Arab Emirates; Lifestyle Intervention; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Behavioral Lifestyle Intervention (3 health centers): In addition to usual care in the health center, the intervention included individual counseling and group education on nutrition and physical activity.
  Interventions: Behavioral: Behavioral Lifestyle Intervention
- Control (Active Comparator): Control (4 health centers): Patients received usual care including education as part of the diabetes management from their healthcare professionals (physicians and nurses), normally every 2-3 months. Visits with the health center dietitian were arranged as per physician referral.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Behavioral Lifestyle Intervention — In addition to usual care in the health center, the intervention included 7 visits with the health center dietitian for individual nutrition counseling, invitation for group nutrition education (5 sessions), individual counseling for physical activity, invitation for a 6-weekly structured group physical activity, DVD on physical activity to perform physical activity at home.
  Arms: Intervention
Behavioral: Usual Care — Patients received usual care including education as part of the diabetes management from their healthcare professionals (physicians and nurses), normally every 2-3 months. Visits with the health center dietitian were arranged as per physician referral.
  Arms: Control

SUMMARY:
The "Skills for Change" Diabetes Nutrition Education Program was a one-year, community-based conducted in Ambulatory Health Care Services health centers in Al Ain. The project involved nutrition education to improve blood glucose control, diet and physical activity levels of Emirati adults with type 2 diabetes.

DETAILED DESCRIPTION:
Despite the high prevalence of diabetes and its complications in the UAE, very few diabetes education intervention studies have been conducted in a representative population in the country. The Skills for Change Program was a one-year, community-based, cluster randomized study involving Emirati adults with type 2 diabetes. We implemented a behavioral lifestyle intervention to improve glycemic control, food choices, and physical activity levels and to decrease sedentarity. The project was culturally adapted to Emirati adults with type 2 diabetes and was driven by theoretical principles of behavior change and education to enhance intervention effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* United Arab Emirates national
* Type 2 diabetes
* Adults: Male and female
* Age: 20-70 years
* Attending one of the 7 health centers in Al Ain managed by the Ambulatory Healthcare Services.

Exclusion Criteria:

* Type 1 diabetes
* Age >70 Years
* Medical conditions that prevent active participation in the program, based on recommendation of the attending physicians
* Participating in other nutrition intervention programs

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2011-11-20 (Actual); Primary Completion 2013-11-28 (Actual); Study Completion 2013-12-24 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 12 months

SECONDARY OUTCOMES:
Change in Total Cholesterol, LDL, HDL and Triglycerides | 12 months
Change in Dietary Intake (Total Calories, Saturated Fat, Cholesterol, Dietary Fiber and Sodium) | 12 months
  Dietary intake was assessed using 24 hour recall with USDA Multiple Pass Method
Change in Physical Activity (total METs and total duration) | 12 months
  Physical Activity was assessed using International Physical Activity Questionnaire Short Form.
Change in Sitting time (minutes) | 12 months
  Sitting time was assessed using International Physical Activity Questionnaire Short Form.
Change in Weight | 12 months
Change in BMI | 12 months
Change in Nutrition Knowledge | 12 months
  Questionnaire was used to assess knowledge of food sources of carbohydrates and dietary fiber
Change in Diabetes Treatment Satisfaction Score | 12 months
  Diabetes Treatment Satisfaction Questionnaire (Bradley,C) was used

CONTACTS AND LOCATIONS:
Overall Officials: Habiba I. Ali, PhD, RD,CDE, Principal Investigator — United Arab Emirates University
Locations (1):
- Ambulatory Healthcare Services, SEHA, Al Ain City, United Arab Emirates

REFERENCES:
- [Derived] Ali HI, Al Ketbi LB, Platat C, Abdl El Baki H, Elmi F, Ibrahim W, Zoubeidi T, Al Dhaheri AS, Cheikh Ismail L, Tariq MNM, Souka U, Yasin J, Stojanovska L. Impact of Skills for Change Program on metabolic control, diet and physical activity levels in adults with type 2 diabetes: A cluster randomized trial. PLoS One. 2024 May 31;19(5):e0304639. doi: 10.1371/journal.pone.0304639. eCollection 2024. PMID 38820345